CLINICAL TRIAL: NCT05451004
Title: SPECT-CT Guided ELEctive Contralateral Neck Treatment for Patients With Lateralized Oropharyngeal Cancer. A Phase III Randomized Controlled Trial
Brief Title: SPECT-CT Guided ELEctive Contralateral Neck Treatment for Patients With Lateralized Oropharyngeal Cancer
Acronym: SELECT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: Alliance for Clinical Trials in Oncology (Other); Eastern Cooperative Oncology Group (Network); NRG Oncology (Other); SWOG Cancer Research Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCTG-HN11; CCTG-HN11 (Other: NCI/CTEP); NCI-2022-04496 (Other: NCI CTRP)
Record Dates: First submitted 2022-06-30; First posted 2022-07-11 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-05

CONDITIONS: Oropharyngeal Cancer
MeSH Terms: conditions — Oropharyngeal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Lympathic Mapping with SPECT-CT guided Radiotherapy (Experimental)
  Interventions: Other: Lymphatic Mapping with SPECT-CT
- Bilateral Neck Radiotherapy (Active Comparator)
  Interventions: Radiation: Ipsilateral and Contralateral Neck

INTERVENTIONS:
Other: Lymphatic Mapping with SPECT-CT — Radiation: Ipsilateral Neck Radiotherapy and SPECT-CT Guided Contralateral Neck Radiotherapy
  Arms: Lympathic Mapping with SPECT-CT guided Radiotherapy
Radiation: Ipsilateral and Contralateral Neck — Radiotherapy
  Arms: Bilateral Neck Radiotherapy

SUMMARY:
This study is being done to answer the following question:

Is the chance of cancer spreading or returning the same if radiotherapy to the neck is guided, by using a special imaging study called lymph node mapping (lymphatic mapping) Single Photon Emission Computed Tomography (SPECT-CT), compared to the usual treatment when radiotherapy is given to both sides of the neck?

DETAILED DESCRIPTION:
This study is being conducted in order to find out if this approach is as good as the usual approach in controlling the cancer and has fewer side effects and better quality of life. The usual approach for patients who are not in a study is treatment which includes radiotherapy to the tumour and to both sides of the neck to decrease the risk of spread or recurrence of the cancer

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathologically proven diagnosis of lateralized OPC (tonsil, tongue base, soft palate, or pharyngeal wall) not involving or crossing midline.
* HPV positive or negative (by p16 immunohistochemistry).
* Clinical stage T1-3 M0 (UICC/AJCC TNM 8th Edition). Nodal involvement may include no nodes or single or multiple ipsilateral lymph nodes (largest ≤6cm in maximum diameter)
* Radiological investigations within 8 weeks of registration:

  * CT or MRI of the neck (with head imaging as indicated);
  * PET-CT scan
  * Chest CT scan
* Planned definitive RT or CRT with bilateral neck RT (patients planned for unilateral neck RT are excluded).
* Intent to deliver concurrent chemotherapy or not must be known at the time of randomization. As this is a pragmatic trial, even patients who are not candidates for systemic therapy will be eligible for participation.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
* Willing to complete the quality of life and/or health utility questionnaire, if sufficiently fluent in available language(s).
* Informed consent prior to registration
* Accessible for treatment and follow-up.
* Commencement of definitive RT within 28 days (+ 14 days) of randomization.
* Injection procedure for lymphatic mapping may be performed in the nuclear medicine, ambulatory clinic, or operating room setting
* Women/men of childbearing potential must have agreed to use a highly effective contraceptive method
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Patient must consent to provision of, and investigator(s) must confirm location and commitment to obtain a representation of formalin fixed paraffin block of non-cytology tumour tissue in order that the specific correlative marker assays

Exclusion Criteria:

* T1-T2 cancers isolated to the tonsil fossa (i.e. without any soft palate, tongue base, posterior pharyngeal wall or posterior tonsil pillar involvement) with no involved lymph nodes or with a single ipsilateral node < 3 cm without extranodal extension.
* Tonsil or tongue base primary cancer who have previously undergone diagnostic palatine or lingual tonsillectomy with either complete excision or with no clinically apparent residual disease
* Previous head and neck cancer or multiple synchronous primary head and neck cancers
* Previous induction or neo-adjuvant chemotherapy.
* Previous radiation therapy to the head and neck or comprehensive neck dissection of at least 3 levels on either side (due to potential for disrupted lymphatic channels and drainage pathways). Patients who have had excisional biopsies of involved lymph nodes are eligible
* Radiotracer allergy
* Severe, active co-morbidity including any of the following:

  * Chronic Obstructive Pulmonary Disease or other pulmonary illness requiring hospitalization within 30 days of registration
  * Unstable angina and/or congestive heart failure requiring hospitalization within the 30 days of registration
  * Acute myocardial infarction within 30 days of study registration
  * Diseases precluding RT (e.g. scleroderma)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 510 (Estimated)
Dates: Start 2023-02-10 (Actual); Primary Completion 2030-08-30 (Estimated); Study Completion 2031-08-30 (Estimated)

PRIMARY OUTCOMES:
Disease-free Survival | 8 years

SECONDARY OUTCOMES:
Quality of Life using M.D. Anderson Dysphagia Inventory (MDADI) | 8 years
  Possible range of scores between 0 and 100 (higher scores indicating better swallowing and lower score indicating poor swallowing).
Xerostomia-related Quality of Life using Xerostomia Questionnaire (XQ) | 8 years
  Clinically meaningful worsening of xerostomia (10 units on XQ) from baseline to 12 months post RT
Isolated contralateral neck failure (iCNF) | 8 years
Overall Survival (OS) | 8 years
Logo-regional Failure (LRF) | 8 years
Distant Metastases (DM) | 8 years
Incidence and Severity of Radiation-related Toxicities | 8 years
Patient-Reported Toxicities using PRO CTCAE | 8 years
Gastrostomy Tube Usage | 8 years
Resource Utilization | 8 years
Lost Productivity | 8 years
  Healthcare system and societal resources will be quantified over the course of the trial to generate utilization information by patient in each study arm. We will generate an average cost per study subject by treatment arm for an overall mean cost per study arm
Financial Toxicity [Financial Index of Toxicity (FIT)] | 8 years
Health Utilities using EQ-5D | 8 years

CONTACTS AND LOCATIONS:
Overall Officials: John R de Almeida, Study Chair — University Health Network, Princess Margaret Hospital, Toronto ON Canada; Ali Hosni, Study Chair — University Health Network, Princess Margaret Hospital, Toronto ON Canada
Locations (33):
- United States (25):
  - City of Hope Corona, Corona, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Moffitt Cancer Center-International Plaza, Tampa, Florida
  - Moffitt Cancer Center - McKinley Campus, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - University of Michigan - Brighton Center for Specialty Care, Brighton, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - MU Health - University Hospital/Ellis Fischel Cancer Center, Columbia, Missouri
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Providence Portland Medical Center, Portland, Oregon
  - MD Anderson in The Woodlands, Conroe, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - MD Anderson West Houston, Houston, Texas
  - MD Anderson League City, League City, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
- Canada (8):
  - BCCA-Vancouver Cancer Centre, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Health Sciences North, Greater Sudbury, Ontario
  - Odette Cancer Centre- Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario
  - CHUM - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke-Fleurimont, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No
Based on CCTG Policy